CLINICAL TRIAL: NCT06078046
Title: MOVIN' CARE for PD: A Project on Community Awareness, Rehabilitation and Empowerment for Parkinson's Disease (Mind-body Interventions)
Brief Title: MOVIN' CARE for PD (Mind-body Interventions)
Acronym: jcpdmcI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Society for Rehabilitation (Other); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA230262I
Record Dates: First submitted 2023-09-21; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Mind-Body Therapies

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Due to the nature of this trial, neither the staff, participants nor care provider can be masked to allocation. The data analyst will be blinded after study completion by having the intervention group information coded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful yoga intervention (Experimental): The intervention, comprising six 90-minute sessions, will be delivered by a trained mindful yoga instructor in group format. The intervention is based on our previously tested mindfulness yoga programme for people with PD (31). Following a universal Hatha Yoga practice, the session comprises mindfulness practice of yoga sequence, breathing exercise, and guided meditation. Both face-to-face and home-based online modes of delivery are available.
  Interventions: Behavioral: Mind-body interventions
- Arts-based therapy intervention (Experimental): Participants in the six 90-minute sessions in this intervention will be engaged in art-making processes through multiple art modalities such as visual arts, dance/ movement, music, drama, and creative writing. Each section is usually structured with Filling-in - greetings and check-in, Bridging - warm-up, Decentering - arts making and appreciation, Harvesting - sharing and response, and Closure. Both face- to-face and home-based online modes of delivery are available.
  Interventions: Behavioral: Mind-body interventions

INTERVENTIONS:
Behavioral: Mind-body interventions — Parallel randomized controlled trial

SUMMARY:
The goal of this intervention study is to investigate the effectiveness of two mind-body interventions - yoga, and arts-based approaches in improving the psycho-social-spiritual well-being among PD patients. The hypotheses include:

H1: Yoga and arts-based interventions will significantly improve the psycho-social-spiritual well-being among PD patients H2: Yoga and arts-based interventions will significantly alleviate or maintain PD-related symptoms and severity levels H3: There is no significant difference between the effectiveness of yoga and arts-based interventions on psycho-social-spiritual well-being among PD patients

Eligible individuals will be invited to a baseline assessment followed by a randomization to the two intervention groups. A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment, to investigate the immediate and long-term effects.

DETAILED DESCRIPTION:
Parkinson's disease (PD), the second most common neurodegenerative disease, usually results in physical deterioration, as well as a spectrum of psychosocial sequels that could bring various challenges on one's daily lives. Patients experience common motor symptoms, including tremor, rigidity, bradykinesia, and postural instability, in parallel with psychosocial stressors (i.e., non- motor symptoms NMS), such as sleep disturbance, cognitive deficits, gastrointestinal symptoms, dopaminergic drug-induced behaviors (e.g., hallucination, impulse control issues) and mood disturbance (e.g., depression, anxiety). While 21% of individuals struggling with the disease reported at least one of these psychosocial symptoms within the initial stage of the disease, they are generally at risk for increased emotional distress, cognitive declines, and elevated stress hormone (cortisol) levels.

Both motor and non-motor symptoms of Parkinson's disease could affect the quality of life of individuals and that of their caregivers. A cross-sectional study conducted by our research team has explored the symptom burden and support care needs in people with PD across East and Southern Asia (n=186), revealing significant unmet needs among Hong Kong PD patients regarding their psychosocial-spiritual concerns. In particular, they experience significant, moderate palliative care needs at the early to middle course of the illness. The extent of unmet support care needs among patients with mild to moderate PD is as great as that among patients with other chronic health conditions, such as advanced cancer, late-stage lung cancer, stage 4/5 chronic obstructive pulmonary disease and late stage chronic kidney disease. The visible and unpredictable symptoms of a distorted body (e.g., tremor and gait dysfunction) and the suppressed expressions due to having a masked face, reduced voice and slurred speech often results in difficulty seeking help and stigmatization of the disease.

Despite the tremendous influences and common occurrence of NMS, they are surprisingly under- recognized in clinical practice because of the lack of spontaneous verbal complaints by the patients, as well as the lack of systematic questioning by healthcare professionals. A qualitative exploration of the illness experience of local PD patients highlighted the importance and urgent need for holistic PD interventions that emphasizes on early identification and preventive measures of individual who are at risk for PD patients, alleviation of the effects of the psychological sequels to PD patients, as well as the reduction of stigma and promotion of community support towards PD.

The study adopts a 2-arm randomized controlled design, aiming to investigate the effectiveness of two mind-body interventions - yoga, and arts-based approaches in improving the psycho-social-spiritual well-being among PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are diagnosed with idiopathic, mild-to-advance PD as indicated by Hoehn and Yahr Scale (19) Stage I to IV (those with unilateral/bilateral symptoms, with/without postural instability who are able to walk at least 3 meters or stand unassisted);
* aged 18 or above;
* able to give written informed consent;
* able to access to the internet and smartphone/ tablet/ laptop will be included; and
* able to comprehend Chinese will be included.

Exclusion Criteria:

* participants have significant cognitive impairment as indicated by the Abbreviated Mental Test lower than 6 significant
* participants have been regularly engaged in regular instructor-led mind-body exercise (e.g., Taichi) or arts-based therapies (>2 times per week) in the past 3 months
* currently participating in any other behavioral or pharmacological trial
* participants have other contraindication(s) that may limit their full participation (e.g. severe hearing or vision impairment, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Change of Perceived stress level | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Perceived Stress Scale (PSS) uses a five-point Likert scale to measure the perceived stress level. The 10 items in the scale can be divided into two subscales, measuring the perceived helplessness, and inadequacy of self-efficacy. The scale ranges from 0-40, with a high score indicates a high perceived stress level. The Cronbach's α of the validated Chinese version of the scale is 0.85.
Change of overall Quality of Life assessed by the WHOQOL-BREF | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Overall quality of life will be measured by the WHOQOL-BREF. It will measure the four dimensions of quality of life, including physical health, psychological health, social relationships, and environment. The scale consists of 26 items and uses a five-point Likert scale. The higher the score, the better the quality of life. The Cronbach's α of the subscales ranges from 0.73-0.82.
Change of Quality of Life specified to Parkinson's Disease assessed by the PDQ-8 | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  The validated Chinese version of Parkinson's Disease Questionnaire-8 consists of 8-items and it captures PD-related health-related quality of life (HRQOL) in eight domains, including mobility, activities of daily living, emotional wellbeing, social support, communication, cognition, body discomfort and stigma. A high score indicates worse HRQOL. Cronbach's α is 0.80.
Change of PD-related symptoms | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  PD-related symptoms will be measured by the validated Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS- UPDRS)(Chinese) Part I to IV [13]. The four dimensions measured by the scale include (i) non-motor experiences of daily living, (ii) motor experiences of daily living, (iii) severity of motor symptoms, and (iv) motor complications. High scores indicate great disease severity. Cronbach's α are 0.79-0.94. In addition, Mon4t (by Montfort Brain
  Monitor, Tel-Aviv, Israel) is a mobile application that evaluates PD-related motor symptoms of participants. It is commonly used for tasks including timed-up-and-go, finger tapping, measuring resting tremor and postural tremor.
Change of self-compassion | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Self-compassion will be measured by the 12-items Self-compassion Scale(SCS). Using a five-points Likert scale, it explores the six dimensions of self-compassion: self- kindness, self-judgment, common humanity, isolation, mindfulness, and over-identified. The total score ranges from 0-60 and will be computed into a mean score (range from 1-5) for analysis. High capacity for self-compassion is reflected by a high score. Cronbach's α is 0.64 for the Chinese version.

SECONDARY OUTCOMES:
Change of self-efficacy assessed by SEMCD | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Self-efficacy will be measured by the Chinese version of Self-efficacy to Manage Chronic Disease Scale (SEMCD). The six-item scale measures the confidence of doing certain activities among people with chronic disease on a 10-point Likert scale. The mean score of the six items is used to reflect the level of self-efficacy, which ranges from 1 to 10. A high score indicates high self-efficacy. Cronbach's α is 0.88.
Change of perceived social support | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Perceived social support will be measured by the adopted version of Duke-UNC Functional Social Support Questionnaire (SSS). On a five-point Likert scale, it measures the perceived supportiveness of other people (e.g., family members, friends, relatives, co-workers, etc.) from the respondent's point of view. The eight items reflect three types of social support: emotional, instrumental, and informational. The scale uses the average score of all items, thus the total mean score ranges from 1 to 5. A higher score indicates greater social support. The Chinese version has Cronbach's α of 0.91.
Change of Constipation severity | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Constipation severity will be measured by the 16-item Chinese version of the Constipation severity instrument (CSI) (Cronbach's α is 0.93-0.95). It consists of three subscales, namely the obstructive defecation, colonic inertia, and pain. The higher the score, the higher the constipation severity (total scores 0-78).
Change of Bowel habits | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Bowel habits will be measured by a self-reported 7-day bowel diary.
Change of Gut microbiota composition | A repeated outcome measure will be conducted at baseline (prior to randomization) (T0), 3-month (T1), 6-month (T2), 9-month (T3) follow-up after baseline assessment
  Fresh stool samples will be collected to investigate participants' gut microbiota composition. Shotgun metagenomics sequencing of the fecal samples will be conducted using the DNBseqTM sequencing platform with a 100 bp paired-end protocol by BGI Tech Solutions (Hong Kong) Co., Ltd. The microbiota composition will be documented by the MetaPhlan3.
User's satisfaction | 3-month (T1)
  User's satisfaction of the intervention will be measured by 11 items on a five- points Likert scale. The scale will be used to understand the participant's satisfaction and perceived effectiveness of the preventive intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rainbow T.H. Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- 2/F., The Hong Kong Jockey Club Building for Interdisciplinary Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No